CLINICAL TRIAL: NCT03135457
Title: A Cross-over Randomized Controlled Trial; Pulmonary Edema Detection After Fluid Loading With Blood Versus Saline in Patients After CABG
Brief Title: TACO Crossover TRIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, A.P.J. Vlaar, MD PhD MBA, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NL59191.018.16
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Transfusion-associated Circulatory Overload; Blood Transfusion Reaction
MeSH Terms: conditions — Transfusion Reaction

STUDY DESIGN:
Intervention Model Description: Open-label, prospective cross-over randomized controlled trial.
Who Masked: Participant, Care Provider
Masking Description: Masking of investigator is not possible due to nature of intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Other): Patients will receive infusion of 300mL saline with a subsequent autologous Red Blood Cells (RBC) transfusion of 300 mL at a rate of 10mL/min
  Interventions: Procedure: Autologous RBC transfusion; Procedure: Saline transfusion
- Group B (Other): Patients will receive infusion of 300mL autologous RBC with a subsequent saline transfusion of 300 mL at a rate of 10mL/min
  Interventions: Procedure: Autologous RBC transfusion; Procedure: Saline transfusion

INTERVENTIONS:
Procedure: Autologous RBC transfusion — Autologous RBC transfusion 300ml 10 ml/min
Procedure: Saline transfusion — Saline transfusion 300ml 10ml/min

SUMMARY:
This is an open-label, prospective crossover randomized controlled trial to investigate wether TACO is solely hydrostatic pressure overload or arises from a combination of hydrostatic pressure overload and capillary leakage, by investigating the difference in change in static pressure parameters (PCWP), dynamic volume parameters (PICCO) as indirect measurements of volume status and capillary leakage after autologous transfusion or saline infusion. The investigators will estimate effective circulating volume following autologous transfusion or saline infusion. Furthermore, the investigators will investigate the effect of fluid loading on the microcirculation.

DETAILED DESCRIPTION:
Coronary arterial bypass grafting surgery patients with reduced left ventricular function will be allocated to either infusion of 300mL saline with a subsequent autologous RBC (cell saver) transfusion of 300 mL at a rate of 10mL/min, or the same in the reversed order. Prior to start of the intervention, 15 minutes following start of infusion and a the end of infusion, the investigators will measure right-ventricular pressure and wedge pressure (PCWP), as well as extravascular lung water index (EVLWI) and CO estimation through PICCO® and Pulmonary Artery Catheter. The investigators will identify fluid responsiveness by performing a passive leg raise test (PLR). The investigators aim to measure total vessel density (TVD), perfused vessel density (PVD), proportion of perfused vessels (PPV), microvascular flow index (MFI), and blood vessel diameters (Øbv) from the oral microcirculation by CytoCam microscope system. The investigators will estimate the effective circulating blood and plasma volume through dilutional infusion of indocyanine green prior to initial infusion, between and at the end of subsequent infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Elective (non-redo) coronary arterial bypass grafting surgery
3. Reduced left ventricular ejection fraction (<55%)
4. Transfusion of autologous blood (cell saver blood, 300ml, HCT60%, 30min)
5. Informed consent

Exclusion Criteria:

1. Patients with no indication for autologous RBC transfusion
2. Patients with pulmonary hypertension, congenital heart disease, mitral or tricuspid valve disease.
3. Contraindications for PAC placement; coagulopathy, bundle branch block, defibrillator or pacemaker (risk of displacement). External pacemaker placed during surgery is no exclusion criterium.
4. Patients for acute, non-elective surgery
5. Chronic kidney disease stage 4 or higher (eGFR < 30)
6. Massive transfusion
7. Previous randomization in the current trial
8. Postoperative ongoing bleeding
9. Bypass duration > 2 hours
10. Infusion of high dose corticosteroids
11. Hemodynamic instability with a mean arterial pressure (MAP) < 60 mmHg, central venous pressure > 20 mmHg or dependence on high dosages of inotropic drugs after admittance to the ICU
12. Severe arrhythmias
13. Development of severe pulmonary edema during infusion of autologous blood or saline.
14. Elevated liver enzymes
15. Iodine allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Hydrostatic pressure overload | 1 hour
  Hydrostatic pressure overload defined as delta pulmonary capillary wedge pressure

SECONDARY OUTCOMES:
Capillary leakage | 1 hour
  Capillary leakage defined as delta extra vascular lung water index
Cardiac output | 1 hour
  Volume overload measured by cardiac output
Mean arterial pressure | 1 hour
  Volume overload measured by mean arterial pressure
Pulse pressure variation | 1 hour
  Volume overload measured by pulse pressure variation
Stroke volume variation | 1 hour
  Volume overload measured by stroke volume variation
Extra vascular lung water index | 1 hour
  Volume overload measured by extra vascular lung water index
Systemic vascular resistance | 1 hour
  Volume overload measured by systemic vascular resistance
Colloid osmotic pressure | 1 hour
  Colloid osmotic pressure measured by membrane colloid osmometer
Estimated circulating volume | 1 hour
  Estimated circulating blood volume measured by indocyanine green
Estimated circulating volume | 1 hour
  Estimated circulating plasma volume measured by indocyanine green
Microcirculation | 1 hour
  Total vessel density in the sublingual microcirculation measured by Cytocam
Microcirculation | 1 hour
  Perfused vessel density in the sublingual microcirculation measured by Cytocam
Microcirculation | 1 hour
  Proportion of perfused vessels in the sublingual microcirculation measured by Cytocam
Microcirculation | 1 hour
  Microvascular flow index in the sublingual microcirculation measured by Cytocam
Microcirculation | 1 hour
  Blood vessel diameters in the sublingual microcirculation measured by Cytocam
Fluid responsiveness | 1 hour
  Fluid responsiveness defined by Passive Leg Raise test (increase in cardiac output > 10%)
TACO | 6 hours
  Transfusion associated circulatory overload criteria 6 hours after infusion of autologous blood transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Vlaar, MD PhD MBA, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam
Locations (1):
- Academisch Medisch Centrum - Universiteit van Amsterdam, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Delaney M, Wendel S, Bercovitz RS, Cid J, Cohn C, Dunbar NM, Apelseth TO, Popovsky M, Stanworth SJ, Tinmouth A, Van De Watering L, Waters JH, Yazer M, Ziman A; Biomedical Excellence for Safer Transfusion (BEST) Collaborative. Transfusion reactions: prevention, diagnosis, and treatment. Lancet. 2016 Dec 3;388(10061):2825-2836. doi: 10.1016/S0140-6736(15)01313-6. Epub 2016 Apr 12. PMID 27083327
- [Derived] Radford M, Estcourt LJ, Sirotich E, Pitre T, Britto J, Watson M, Brunskill SJ, Fergusson DA, Doree C, Arnold DM. Restrictive versus liberal red blood cell transfusion strategies for people with haematological malignancies treated with intensive chemotherapy or radiotherapy, or both, with or without haematopoietic stem cell support. Cochrane Database Syst Rev. 2024 May 23;5(5):CD011305. doi: 10.1002/14651858.CD011305.pub3. PMID 38780066